CLINICAL TRIAL: NCT04414267
Title: A Randomized Clinical Trial for Enhanced Trained Immune Responses Through Bacillus Calmette-Guérin Vaccination to Prevent Infections by COVID-19: The ACTIVATE II Trial
Brief Title: Bacillus Calmette-guérin Vaccination to Prevent COVID-19
Acronym: ACTIVATEII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Activate II; 2020-002448-21 (EudraCT Number)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: COVID-19; Virus Diseases; Corona Virus Infection; Coronary Heart Disease; Chronic Obstructive Pulmonary Disease
Keywords: COVID-19; SARS-CoV-2; Vaccination; Bacillus Calmette-Guérin vaccination
MeSH Terms: conditions — COVID-19; Virus Diseases; Coronavirus Infections; Coronary Disease; Pulmonary Disease, Chronic Obstructive | interventions — BCG Vaccine; Freeze Drying; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients vaccinated with placebo or BCG
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG vaccine (Experimental): One intradermal injection of 0.1ml of BCG (BCG vaccine Moscow strain 361-1; Serum Institute of India Pvt. Ltd)
  Interventions: Biological: BCG vaccine
- Placebo (Placebo Comparator): One intradermal injection of 0.1ml of sodium chloride 0.9%
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BCG vaccine — Patients susceptible to SARS-CoV-2 infection will be vaccinated with one intradermal injection of 0.1ml of BCG vaccine
  Other Names: BCG Vaccine (Freeze Dried)
  Arms: BCG vaccine
Biological: Placebo — Patients susceptible to SARS-CoV-2 infection will be vaccinated with one intradermal injection of 0.1ml of sodium chloride 0.9%
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Based on findings of the interim analysis of the ACTIVATE study showing 53% decrease of the incidence of all new infections with BCG vaccination, a new trial is designed aiming to validate if BCG can protect against COVID-19 (Corona Virus Disease-19).The aim of the study is to demonstrate in a double-blind, placebo-controlled approach if vaccination of participants susceptible to COVID-19 with BCG vaccine may modulate their disease susceptibility for COVID-19. This will be validated using both clinical and immunological criteria. At the same time, a sub-study will be conducted and the mechanism of benefit from BCG vaccination by assessing its effect on vascular endothelial function and mononuclear blood cells will be studied

DETAILED DESCRIPTION:
Infection by the novel SARS-CoV-2 virus (also known as COVID-19) has tremendous social impact. Most of Western societies are at major or part lock-down whatever brings unpredictable financial and societal consequences. The urgent need for the reversal of this situation can only be met through the generation of an immune defence shield to protect the society from COVID-19. Many efforts for the development of a vaccine are under way without any specific outcome so for.

The stimulation of trained immune responses seems the only alternative to bridge the gap from the turn-on of the society until the entrance of a specific vaccine in the market. Trained immunity stands for the non-specific raise of defense shield for severe infections coming once tissue macrophages recognize a universal pathogen. The concept was successfully tested in healthy volunteers that were vaccinated with placebo or BCG (Bacillus Calmette-Guérin) vaccine. These volunteers were injected 14 days latter a tri-valent influenza A vaccine. Volunteers previously vaccinated by BCG developed significantly greater titers against hemagglutinin A of the influenza A virus whereas their circulating monocytes were more potent for the production of interferon-gamma.

It is proposed that this BCG vaccination triggering trained immune responses may play a role of protection against the COVID-19 pandemic. A solid background on this rationale came recently from the interim analysis of the ACTIVATE trial. ACTIVATE (A randomized Clinical trial for enhanced Trained Immune responses through Bacillus Calmette-Guérin VAccination to prevenT infections of the Elderly) was a prospective randomized open-label controlled trial conducted among patients hospitalized at the 4th Department of Internal Medicine of ATTIKON University General Hospital in Greece. The protocol was approved by the National Ethics Committee of Greece and the National Organization for Medicine of Greece (EudraCT number, 2017-000596-87; ClinicalTrials.gov NCT03296423). The trial is conducted and funded by the Hellenic Institute for the Study of Sepsis. In this trial hospitalized elderly patients were vaccinated on the day of hospital discharge with single doses of placebo or BCG. Every patient is under follow-up for 12 months. The last visit of the last patient is scheduled for August 2020. An interim analysis took place on April 29th 2020 by an independent committee of experts. The full interim analysis focused on the study primary endpoint that was the comparative time to a new infection between the two groups of treatment. Infections counting against this primary endpoint were respiratory or viral infections necessitating medical treatment, community-acquired pneumonias, hospital-acquired pneumonias, intraabdominal infections, urinary tract infections, soft tissue infections and bloodstream infections. Analysis revealed 53% decrease of the incidence of new infections in the BCG group compared to the placebo group. This decrease reached 80% for all respiratory tract infections. Multivariate analysis showed that most of benefit was for patients with coronary heart disease (CHD) and chronic obstructive pulmonary disease (COPD). This interim analysis clearly enhances the concept that BCG can be protective against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female
3. Age more than or equal to 50 years based on the precise date of birth. Female participants are allowed on the premise that they are post-menopausal.
4. History of at least one of the following:

   1. coronary heart disease;
   2. chronic obstructive pulmonary disease;
   3. Charlson's comorbidity index (CCI) more than 3
5. Negative serum testing for immunoglobulin G and M against SARS-CoV-2
6. Skin tuberculin test diameter less than 10mm

Exclusion Criteria:

* Deny to written informed consent
* Age less than 50 years
* Known infection by the Human Immunodeficiency Virus-1 (HIV-1)
* Severely immunocompromised patients. This exclusion category comprises:

  * History of congenital immunodeficiency
  * History of solid organ transplantation
  * History of bone marrow transplantation
  * Intake of chemotherapy the last two months
  * Intake of radiotherapy the last two months
  * Active hematological or solid tumor malignancy
  * History of any anti-cytokine therapies
  * History of oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than the last 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Positive for the respiratory questionnaire consisted of questions concerning the appearance of symptoms possibly, probably and/or definitively related to COVID-19 on visit 3. | Visit 3 (90 +/- 5 days)
  This is set on visit 3 (90 ± 5 days from the date of visit 1). The two groups of vaccination are compared for the primary endpoints which is composite. Patients who meet any of the following will be considered to meet the primary endpoint:
  * Positive for the respiratory questionnaire endpoint when at least one of the following combination is met either at visit 2 and/or at visit 3:
    * One situation definitively related to COVID-19
    * All four questions of symptoms possibly related to COVID-19
    * At least two questions of symptoms possibly related to COVID-19 as well as need for admission at the emergency department of any hospital and/or need for intake of antibiotics
    * At least four questions of symptoms probably related to COVID-19 one of which is "need for admission at the emergency department of any hospital and/or need for intake of antibiotics"
  * Positive IgG or IgM antibodies against SARS-CoV-2

SECONDARY OUTCOMES:
Positive respiratory questionnaire endpoint consisted of questions concerning the appearance of symptoms possibly, probably and/or definitively related to COVID-19 on visit 4 | Visit 4 (135 +/- 5 days)
  The two groups of vaccination are compared for the primary endpoints which is composite (as defined at primary study endpoint) and meet a positive respiratory questionnaire endpoint on visit 4
Positive respiratory questionnaire endpoint consisted of questions concerning the appearance of symptoms possibly, probably and/or definitively related to COVID-19 on visit 5 | Visit 5 (180 +/- 5 days)
  The two groups of vaccination are compared for the primary endpoints which is composite (as defined at primary study endpoint) and meet a positive respiratory questionnaire endpoint (as defined at primary study endpoint) on visit 5
Prevalence of IgG/IgM against SARS-CoV-2 | Screening Visit and Visit 3 (90 +/- 5 days)
  Prevalence of IgG/IgM against SARS-CoV-2 will be measured among the patients who failed the eligibility procedure and the patients that were eligible and were enrolled
Analysis of each of the components of the respiratory questionnaire consisted of questions concerning the appearance of symptoms possibly, probably and/or definitively related to COVID-19. | Visit 2 (45 +/- 5 days), Visit 3 (90 +/- 5 days), Visit 4 (135 +/- 5 days), Visit 5 (180 +/- 5 days)
  Itemized analysis of each of the components of the respiratory questionnaire on each study visit
The impact of new cardiovascular events between the two study groups | Visit 2 (45 +/- 5 days), Visit 3 (90 +/- 5 days), Visit 4 (135 +/- 5 days), Visit 5 (180 +/- 5 days)
  The impact of new cardiovascular events between the two study groups (placebo and BCG) will be analyzed, though the collection of any cardiovascular events occured to the enrolled patients.
Differences in repeated measurements of angiometric parameters (arterial hardness) between the two sub-study groups in Visit 3 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days)
  Differences in repeated measurements of arterial stiffness in visit 3 between the two sub-study groups (placebo or BCG) will be analyzed through the speed of the pulse wave velocity. Pulse wave velocity is measured in m/sec.
Differences in repeated measurements of angiometric parameters (central arterial pressures and reflected waves) between the two sub-study groups in Visit 3 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days)
  Differences in repeated measurements of central arterial pressures and reflected waves in visit 3 between the two sub-study groups (placebo or BCG) will be measured non-invasively by pulse wave analysis. Central arterial pressure is measured in mmHg.
Differences in repeated measurements of angiometric parameters (endothelial function) between the two sub-study groups in Visit 3 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days)
  Differences in repeated measurements of endothelial function in visit 3 between the two sub-study groups (placebo or BCG) will be measured by ultrasound measurement of endothelium-dependent flow-mediated dilatation and by nitrate-mediated dialatation. Endothelial function will be assessed by Flow Mediated Dilatation (FMD). Endothelium-dependent: diameter of the artery prior and after temporary ischemia in is measured in mm, nitrate-mediated: diameter of the artery prior and after nitrate administration is measured in mm
Differences in repeated measurements of angiometric parameters (thickness of the medial carotid sheath) between the two sub-study groups in Visit 3 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days)
  Differences in repeated measurements of thickness of the medial carotid sheath in visit 3 between the two sub-study groups (placebo or BCG) will be measured by B-mode ultrasound examination. Intima-Media Thickness is measured in mm
Differences in repeated measurements of angiometric parameters (arterial hardness) between the two sub-study groups in Visit 5 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days), Visit 5 (180 +/- 5 days)
  Differences in repeated measurements of arterial stiffness in visit 5 between the two sub-study groups (placebo or BCG) will be analyzed through the speed of the pulse wave velocity. Pulse wave velocity is measured in m/sec.
Differences in repeated measurements of angiometric parameters (central arterial pressures and reflected waves) between the two sub-study groups in Visit 5 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days), Visit 5 (180 +/- 5 days)
  Differences in repeated measurements of central arterial pressures and reflected waves in visit 5 between the two sub-study groups (placebo or BCG) will be measured non-invasively by pulse wave analysis. Central arterial pressure is measured in mmHg.
Differences in repeated measurements of angiometric parameters (thickness of the medial carotid sheath) between the two sub-study groups in Visit 5 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days), Visit 5 (180 +/- 5 days)
  Differences in repeated measurements of thickness of the medial carotid sheath in visit 5 between the two sub-study groups (placebo or BCG) will be measured by B-mode ultrasound examination. Intima-Media Thickness is measured in mm
Differences in repeated measurements of angiometric parameters (endothelial function) between the two sub-study groups in Visit 5 | Visit 1 (Day 0), Visit 3 (90 +/- 5 days), Visit 5 (180 +/- 5 days)
  Differences in repeated measurements of endothelial function in visit 5 between the two sub-study groups (placebo or BCG) will be measured by ultrasound measurement of endothelium-dependent flow-mediated dilatation and by nitrate-mediated dialatation. Endothelial function will be assessed by Flow Mediated Dilatation (FMD). Endothelium-dependent: diameter of the artery prior and after temporary ischemia in is measured in mm, nitrate-mediated: diameter of the artery prior and after nitrate administration is measured in mm
Differences in cardiac ultrasound at visit 5 between the two sub-study groups | Visit 1 (Day 0), Visit 3 (90 +/- 5 days), Visit 5 (180 +/- 5 days)
  Differences in cardiac ultrasound at visit 5 between the two sub-study groups (placebo or BCG) will be assessed using standard measurements from 2-D and Doppler echocardiography.
Changes in the release of cytokines from blood mononuclear cells at visit 3 between the two sub-study groups | Visit 1 (Day 0), Visit 3 (90 +/- 5 days)
  Changes in the release of cytokines from blood mononuclear cells at visit 3 between the two sub-study groups (placebo or BCG) will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Papadopoulos, MD, PhD, Principal Investigator — National Kapodistrian University of Athens, Medical School
Locations (15):
- Greece (15):
  - General Hospital of Argolida - Nafplion Unit, Nafplion, Argos
  - 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Alexandroupoli
  - Department of Therapeutics, Alexandra General Hospital, Athens
  - 1st Department of Internal Medicine, General Hospital of Athens G. GENNIMATAS, Athens
  - 2nd University Department of Internal Medicine, IPPOKRATEION General Hospital of Athens, Athens
  - 3rd University Department of Internal Medicine, General Hospital of Chest Diseases of Athens I SOTIRIA, Athens
  - 4th Department of Internal Medicine, "Attikon" University Hospital, National and Kapodistrian University of Athens, Medical School, Athens
  - Department of Pulmonary Medicine- General Hospital of Kerkyra, Corfu
  - General Hospital of Korinthos, Corinth
  - 1st Department of Internal Medicine, General University Hospital of Ioannina, Ioannina
  - Department of Internal Medicine, General Hospital of Karditsa, Karditsa
  - Department of Internal Medicine, Patras University Hospital, Pátrai
  - General Hospital of Ptolemaida MPODOSAKEIO, Ptolemaida
  - 1st Department of Internal Medicine, AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Imathia - Veria Unit, Véria

IPD SHARING:
Plan to Share IPD: No